CLINICAL TRIAL: NCT04123639
Title: Outcomes of Endovascular Treatment of Superficial Femoral Artery In-stent Restenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mark Malak Mahrous, Principal Investigator, Assiut University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 16
Record Dates: First submitted 2019-10-06; First posted 2019-10-11 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: PTA — Percutaneous transluminal angioplasty

SUMMARY:
Lower limb peripheral arterial disease (PAD) is a common, important manifestation of systemic atherosclerosis. Stenosis or occlusions in the superficial femoral artery (SFA) may result in intermittent claudication or even critical ischemia, which may be treated by balloon angioplasty with or without stenting .

Atherosclerotic disease in the femoropopliteal (FP) artery consists of perfusion to the legs and feet. Percutaneous transluminal angioplasty (PTA) has been routinely used to manage FP artery disease and is recommended as an alternative to surgical bypass. Recently, newer endovascular approaches such as covered stent, drug-eluting balloon (DEB), drug-eluting stent (DES), or catheter based atherectomy have been introduced as treatment options for FP artery disease. Nevertheless, FP artery-in stent restenosis (ISR) is still a major challenge with endovascular therapy .

Although the use of peripheral arterial stents brought about a dramatic improvement in patients' clinical and procedural outcomes, the long-term outcome of stent implantation remains significantly constrained by the risk of developing in-stent restenosis (ISR) over time.

Advancements in endovascular stent technology have addressed limitations associated with conventional percutaneous transluminal balloon angioplasty in patients with chronic peripheral arterial disease (PAD) of the lower limbs, such as elastic recoil,residual stenosis and flow-limiting dissection . However, a considerable proportion of patients with PAD treated with stenting will require secondary interventions due to in-stent restenosis (ISR), which is particularly common in long and complex lesions ISR refers to loss of luminal volume from an ingrowth of cells, extracellular matrix, and thrombus within the cylinder of the stented artery and 5-mm margins proximal and distal to the stent. ISR has been reported to occur in 18-40% of patients undergoing stenting in the femoropopliteal segment within the first year of treatment .

The treatment of ISR is one of the major challenges in endovascular therapy for PAD. The treatment options for ISR include standard balloon angioplasty with or without repeat stenting (using bare-metal stents, stent grafts or drug-eluting stents), drug-coated or cutting balloon angioplasty, cryoplasty and directional or laser atherectomy .

ELIGIBILITY:
Inclusion Criteria:

- Patients with PAD undergoing peripheral vascular intervention with SFA in stent stenosis for two years from the start of study and has critical limb ischemia.

Exclusion Criteria:

* Refusal of the patients

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Change number of superficial femoral artery in stent restenosis | 3 years
  Change number of superficial femoral artery in stent restenosis

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No